CLINICAL TRIAL: NCT01775397
Title: A Phase IIIb/IV Randomized, Controlled, Double-blind, Double-dummy, Parallel Group Study to Compare the Efficacy of Fidaxomicin to Vancomycin in the Sustained Clinical Cure of Clostridium Difficile Infection in Adults Receiving Immunosuppressive Therapy
Brief Title: A Post-marketing, Blinded Study to Investigate How Effective Fidaxomicin is Compared to Vancomycin in the Sustained Cure of Clostridium Difficile Infection in Adults That Are Receiving Therapy to Suppress the Immune System
Acronym: FREEDOM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to difficulty in enrollment
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FID-EC-0001; 2012-000531-88 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-25 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Clostridium Difficile
Keywords: Dificid; Infections; Clostridium; Transplantation; Efficacy; Adult; Stem Cells; Fidaxomicin; Difficile; Immunosuppression; Vancomycin
MeSH Terms: conditions — Infections | interventions — Fidaxomicin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fidaxomicin (Experimental): Fidaxomicin with alternating matching placebo
  Interventions: Drug: Fidaxomicin; Drug: Placebo
- Vancomycin (Active Comparator): Participants received 4 doses (1 dose every 6 hours) of oral vancomycin hydrochloride each day for the duration of the 10-day treatment period
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin — capsule
  Other Names: Dificlir®
  Arms: Fidaxomicin
Drug: Vancomycin — capsule
  Other Names: Vancocin®
  Arms: Vancomycin
Drug: Placebo — Capsule
  Arms: Fidaxomicin

SUMMARY:
The primary objective is to compare fidaxomicin versus vancomycin for the sustained clinical cure of Clostridium difficile Infection (CDI) in adult patients receiving immunosuppressive therapy.

DETAILED DESCRIPTION:
On Day 1, subjects with diarrhea defined as having three or more unformed bowel movements or >200 mL of unformed stool (for subjects having rectal collection devices) within 24 hours, confirmed by a rapid CDI test (positive for both toxins A & B and glutamate dehydrogenase) to have CDI will be randomized to receive fidaxomicin or vancomycin (1:1 randomization).

Subjects will be treated with study medication from Day 1 to Day 10. Assessment for clinical cure (Test of Cure [TOC]) will take place 48 - 72 hours after End of Treatment (EOT). Subjects not meeting the definition of clinical cure at TOC will be defined as treatment failures.

A stool sample for evaluation of microbial cure will be taken at TOC on Day 12.

Subjects meeting the criteria for clinical cure at TOC will be monitored for recurrence until 28 days after TOC (Day 40).

Treatment of subjects with recurrence of CDI will be at the

discretion of the Investigator.

Subjects not meeting the criteria for clinical cure at TOC will be followed for safety until Day 40. Further CDI treatment will be at the discretion of the Investigator.

The strain of Clostridium difficile will be determined for all samples.

ELIGIBILITY:
Inclusion Criteria:

* CDI is confirmed by clinical symptoms and rapid CDI test
* Subject has not been treated with medication for CDI within the last 10 days
* Subject is:

  * receiving immunosuppressive therapy (chemotherapy) or is undergoing a stem cell transplant procedure (defined as the time period from the start of conditioning prior to transplant until 6 months after infusion of stem cells) for a hematological malignancy; or
  * receiving immunosuppressive therapy (chemotherapy) for a solid tumor malignancy or following solid organ transplantation; or
  * being treated with immunosuppressive and /or anti-TNF therapy for an auto-immune disease
* Any woman of childbearing potential requires negative serum or urine pregnancy test before entry to the study
* Male and female subjects that are sexually active must agree to practice effective birth control during the study and for 30 days after the end of the study

Exclusion Criteria:

* The subject has experienced more than one previous episode of CDI within the 3 months prior to study inclusion
* Taking or requiring to be treated with prohibited medications
* Unable to take oral study medication
* Female patients that are pregnant, intend to become pregnant or are breastfeeding
* History of ulcerative colitis or Crohn's disease
* History or diagnosis of toxic megacolon or pseudomembranous colitis
* Hypersensitivity to fidaxomicin or any of its components
* Hypersensitivity to vancomycin or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

PRIMARY OUTCOMES:
Sustained clinical cure of CDI at day 26 | Day 26
  Clinical cure is defined as a subject that at TOC no further CDI therapy is required since completion of study medication, and has either:
  * ≤3 unformed bowel movements for two consecutive days
  * ≥50% reduction in the number of unformed bowel movements compared to baseline; or
  * 75% reduction in the volume of liquid stool collected or no longer passing liquid stools (for subjects having rectal collection device)

SECONDARY OUTCOMES:
Clinical Cure of CDI | Day 12
  Clinical cure is defined as a subject that at TOC no further CDI therapy is required since completion of study medication, and has either:
  * ≤3 unformed bowel movements for two consecutive days
  * ≥50% reduction in the number of unformed bowel movements compared to baseline; or
  * 75% reduction in the volume of liquid stool collected or no longer passing liquid stools (for subjects having rectal collection device)
Sustained Clinical Cure of CDI at day 40 | Day 40
  Clinical cure is defined as a subject that at TOC no further CDI therapy is required since completion of study medication, and has either:
  * ≤3 unformed bowel movements for two consecutive days
  * ≥50% reduction in the number of unformed bowel movements compared to baseline; or
  * 75% reduction in the volume of liquid stool collected or no longer passing liquid stools (for subjects having rectal collection device)
Microbial Eradication | Day 12
  Total viable count of clostridium difficile recovered from fecal specimen is below the limit of detection
Resolution of diarrhea | Day 12
  First of two days with <3 bowel movements per day
Use of further CDI therapy required | Between Day 10 and Day 12
Number of unformed stools | Between Day 10 and Day 12
>50% reduction in number of unformed stools compared to baseline | Day 1 to Day 12
Recurrence of CDI | Between Day 1 and Day 40
  After TOC, re-establishment of diarrhea to an extent that is greater than the frequency recorded on the last day of study medication
Time to recurrence of CDI | Between Day 12 and Day 40
  Time elapsing (days) from TOC to confirmed recurrence of CDI

CONTACTS AND LOCATIONS:
Overall Officials: Associate Director Medical Affairs, Study Director — Astellas Pharma Europe Ltd.
Locations (16):
- Univ. Klinik für Innere Medizi, Salzburg, Austria
- Herlev University Hospital, Herlev, Denmark
- France (2):
  - Institut Curie, Paris
  - Hôpital Necker, Paris
- Germany (4):
  - Charité, Berlin
  - Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum, Essen
  - Universitätsklinikum Halle, Halle
- Greece (4):
  - General Hospital of Athens, Athens
  - Laiko General Hospital, Athens
  - University Hospital of Crete, Heraklion
  - Metaxa Anticancer Hospital, Piraeus
- Szpital Specjalistyczny w Brzo, Brzozów, Poland
- Spain (3):
  - H. U. de Bellvitge, Barcelona
  - H.U. Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=345